CLINICAL TRIAL: NCT02343549
Title: A Phase II Study of Optune (NovoTTF) in Combination With Bevacizumab (BEV) and Temozolomide (TMZ) in Patients With Newly Diagnosed Unresectable Glioblastoma (GBM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: closed to accrual due to low accrual
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCI-NEU-NOV-001; 00010270
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2021-09

CONDITIONS: Cancer of Brain and Nervous System
MeSH Terms: conditions — Brain Neoplasms; Neurologic Manifestations | interventions — Bevacizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Planned RT + TMZ + BEV + NovoTTF100A Device (Experimental): Best standard of care radiation therapy (RT, 2 Gy given daily 5 days per week), temozolomide (TMZ, 75 mg/m2 administered daily), and bevacizumab (BEV, 10 mg/kg administered every 2 weeks as an IV infusion) for 6 weeks. After completion of chemoradiation, NovoTTF100A system was initiated, to be worn on average 18 hours or more a day for up to 12 months. The patients also continued with maintenance TMZ/BEV.
  Interventions: Device: NovoTTF100A; Drug: Bevacizumab; Drug: Temozolomide

INTERVENTIONS:
Device: NovoTTF100A
  Other Names: Optune(TM)
Drug: Bevacizumab
  Other Names: Avastin
Drug: Temozolomide
  Other Names: Temodar

SUMMARY:
All patients will complete best standard of care radiation, temozolomide and bevacizumab (6 weeks). Within two weeks of completion of this initial treatment period, study patients will be fitted with the NovoTTF-100A System and treated continuously. They will be treated with TTFields for 12 months for an average of 18 hours per day. The patient may elect to take a treatment break for a total of 3 days per month, for each month and still be in compliance. This will consist of wearing four electrically insulated electrode arrays on the head. The patients will also continue with maintenance temozolomide/ bevacizumab.

DETAILED DESCRIPTION:
This study will be carried out in two stages. The first stage will enroll a cohort of 22 patients. The FDA will review safety data of the first 15 patients during enrollment of the first cohort. Enrollment and interim analysis of the first cohort of patients will be completed within 15 months of study commencement. Upon FDA approval and favorable interim analysis followed by subsequent protocol/consent amendment (as applicable), the second stage will enroll a cohort of 24 patients and will be completed within 15 months of stage 2 commencement. The overall duration of the study is expected to be no longer than 30 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years of age
* Have undergone a brain biopsy via stereotactic or open technique
* Pathological evidence of GBM using WHO classification criteria
* Planned 6 weeks of concurrent chemoradiotherapy post-biopsy concomitant with temozolomide (45-70Gy)
* Karnofsky scale greater than or equal to 70
* Life expectancy at least 3 months
* Baseline hemoglobin of > 8.0 gm/dL (with or without transfusion)
* Adequate coagulation defined as PT and INR < 1.5 times the upper limit of normal
* Signed informed consent
* Able to start bevacizumab at least 2 weeks but no more than 4 weeks from date of biopsy
* Able to tolerate MRI of brain and have measurable disease.
* Participants of childbearing age must use effective contraception for at least 6 months following completion of treatment.

Exclusion Criteria

* Enrolled in another clinical treatment trial
* Pregnant or Breast-feeding
* Any other malignancy aside from localized basal cell or squamous cell carcinoma of the skin
* Significant co-morbidities at baseline which would prevent maintenance temozolomide
* Thrombocytopenia (platelet count < 100 x 103 )
* Neutropenia (absolute neutrophil count < 1.5 x 103 )
* CTC grade 4 non-hematological toxicity (except for alopecia, nausea, vomiting)
* Significant liver function impairment - AST or ALT > 3 times the upper limit of normal
* Total bilirubin> 2 times the upper limit of normal
* Significant renal impairment (serum creatinine> 1.7 mg/dL)
* Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
* Infra-tentorial tumor
* Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea, or reduced level of consciousness)
* History of hypersensitivity reaction to temozolomide or a history of hypersensitivity to DTIC or hydrogel
* Inability to adequately cover treatment area with TTFields (Tumor Treating Fields)
* Inability to wear NovoTTF-100A System for an average of 18 hours per 24 hours
* Currently taking cytotoxic medications, non-steroidal ant-inflammatory drugs (NSAIDS), or enzyme inducing anticonvulsants.
* Currently taking anticoagulants or blood-thinners (Coumadin)
* Subjects meeting any of the following bevacizumab-specific contraindications are ineligible for study entry:
* Inadequately controlled hypertension (defined as systolic blood pressure greater than or equal to 150 and/or diastolic blood pressure > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to study enrollment
* History of hemoptysis (greater than or equal to a half teaspoon of bright red blood per episode) within 1 month prior to study enrollment
* Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure or significant traumatic injury within 28 days prior to 1st bevacizumab infusion or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation within 6 months prior to study enrollment
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria at screening as demonstrated by either urine protein: creatinine (UPC) ratio greater than or equal to 1.0 at screening OR urine dipstick for proteinuria greater than or equal to 2 or more (patients discovered to have greater than or equal to 2 or greater proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate less than or equal to 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-01; Primary Completion 2020-07-11 (Actual); Study Completion 2020-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Sumrall, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Planned RT + TMZ + BEV + NovoTTF100A Device
Started | 13
Completed | 0
Not Completed | 13
Not completed — Death | 11
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Planned RT + TMZ + BEV + NovoTTF100A Device
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 62 [44 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13
Karnofsky Performance Scale [Count of Participants; unit: Participants] — Karnofsky Performance Scale (KPS) classifies level of functional impairment, where 100 indicates normal function/no evidence of disease, while 0 indicates death.
  Participants
    100 - Normal, no complains, no evidence of disease | 1
    90 - Able to carry on normal activity; minor signs or symptoms of disease | 4
    80 - Normal activity with effort; some signs or symptoms of disease | 3
    70 - Cares for self, unable to carry on normal activity or to do active work | 4
    60 - Requires occasional assistance, but is able to care for most of his/her needs | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 12-Month Survival
Description: Twelve-month survival was determined for each subject as a binary variable indicating whether or not the subject was alive at 12 months from initiation of chemoradiation. Determination of this endpoint occurs after the subject has at least 12 months of follow-up, unless they have died sooner.
Time Frame: Evaluated over 12 months
Population: The evaluable population for efficacy includes subjects who receive initial placement of the NovoTTF100A transducer arrays. Note: 4 subjects discontinued study participation prior to device placement but after initiation of RT+TMZ+BEV, and are therefore are excluded from efficacy analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Planned RT + TMZ + BEV + NovoTTF100A Device
Number analyzed (Participants) | 9
Participants | 3
Statistical Analysis 1: Comparison: Planned RT + TMZ + BEV + NovoTTF100A Device; Assuming the true 12-month survival rate is 0.30 under the null hypothesis, then this design will provide 90% power to detect a difference of 0.20 under the alternative hypothesis, assuming a one-sided alpha = 0.10 significance level. A Simon optimal 2-stage design with Stage 1 n=22 and a total of n=46 subjects was determined with the following rejection regions: For n = 22, the rejection region in number of subjects alive at 12 months is 0 - 7, and for n = 46 it is 8 - 17; Test type: Superiority; p = 0.537, Fisher Exact — This p-value is only based on partial enrollment of Stage 1. As enrollment was halted early, this p-value is descriptive in nature and cannot determine the success/failure of the trial; 12-Month Survival Rate = 0.333, 95% CI 2-sided [0.075 to 0.701] — Confidence interval estimated using the Clopper Pearson method

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the duration from the initiation of chemoradiation therapy to the date of death from any cause. Subjects who were alive or lost to follow-up at the time of the analysis were be censored at the last known date they were alive.
Time Frame: From date of treatment start to date of death, or censored as described above; assessed for approximately 5 years
Population: The evaluable population for efficacy includes subjects who receive initial placement of the NovoTTF100A transducer arrays. Note: 4 subjects discontinued study participation prior to device placement, and are therefore are excluded from efficacy analyses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Planned RT + TMZ + BEV + NovoTTF100A Device
Number analyzed (Participants) | 9
months | 9.9 [4.8 to 12.8]
Statistical Analysis 1: Comparison: Planned RT + TMZ + BEV + NovoTTF100A Device; Test type: Other — Estimation Only; Median = 9.9, 95% CI 2-sided [4.8 to 12.8] — The Kaplan Meier method was used to estimate median OS(in months). The Greenwood method was used to estimate confidence limits of median overall survival

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-Free Survival (PFS) is defined as duration of time from initiation of chemoradiation therapy to first occurrence of either progressive disease (PD) or death. PD must be objectively determined as per RANO criteria (Updated Response Assessment Criteria for High Grade Gliomas, where PD is defined as a 25% increase in sum of products of diameters from nadir), where date of PD is date of assessment that identified PD. If subject died without documented PD, date of progression will be date of death. For surviving subjects who do not have documented PD, PFS will be censored at date of last radiologic assessment. For subjects who receive subsequent anti-cancer therapy prior to documented PD, PFS will be censored at the date of last radiologic assessment prior to the commencement of subsequent therapy. Subjects who have an initial PFS event immediately following 2 or more consecutive missed assessments will be censored at date of last assessment prior to missed assessments.
Time Frame: From date of treatment start to date of progression/death, or censored as described above; assessed for approximately 2 years.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Planned RT + TMZ + BEV + NovoTTF100A Device
Number analyzed (Participants) | 9
months | 7.9 [4.8 to 10.4]
Statistical Analysis 1: Comparison: Planned RT + TMZ + BEV + NovoTTF100A Device; Test type: Other — Estimation Only; Median = 7.9, 95% CI 2-sided [4.8 to 10.4] — The Kaplan Meier method was used to estimate median PFS (in months). The Greenwood method was used to estimate confidence limits of median progression free survival

4. Secondary Outcome: Number of Participants With Objective Response
Description: Objective response was determined for each subject as a binary variable indicating whether or not the subject achieved a best overall response of complete response (CR) or partial response (PR) as determined by the Updated Response Assessment Criteria for High Grade Gliomas (RANO; where CR is indicated by disappearance of all target lesions and PR is indicated by >=50% decrease in the sum of products of diameters of target lesions with baseline as reference). Best responses of CR or PR must be confirmed by a subsequent radiologic assessment.
Time Frame: From enrollment to best response while on study treatment; subjects remained on treatment until disease progression or death or unacceptable toxicity (subjects were on treatment for an average of 7 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Planned RT + TMZ + BEV + NovoTTF100A Device
Number analyzed (Participants) | 9
Participants | 3
Statistical Analysis 1: Comparison: Planned RT + TMZ + BEV + NovoTTF100A Device; Test type: Other — Estimation only; Response Rate = 0.333, 95% CI 2-sided [0.075 to 0.701] — Confidence interval estimated using the Clopper Pearson method

5. Secondary Outcome: Number of Participants With Disease Control
Description: Disease control was determined for each subject indicating whether or not they achieved an overall response of stable disease (SD) or better by RANO criteria (where a CR is indicated by disappearance of all target and non target lesions, a PR is indicated by >= 50% decrease in sum of products of diameters of target lesions with baseline as reference, and SD is neither sufficient shrinkage to qualify for PR nor sufficient growth, >=25%, to indicate progression).
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Planned RT + TMZ + BEV + NovoTTF100A Device
Number analyzed (Participants) | 9
Participants | 9
Statistical Analysis 1: Comparison: Planned RT + TMZ + BEV + NovoTTF100A Device; Test type: Other — Estimation only; Disease Control Rate = 1.000, 95% CI 2-sided [0.664 to 1.000]

6. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was measured from the time RANO criteria are met for CR or PR (whichever is first recorded) until the first occurrence of either progressive disease or death. PD must be objectively determined as per RANO criteria (Updated Response Assessment Criteria for High Grade Gliomas, where PD is defined as a 25% increase in sum of products of diameters from nadir), where PD date is assessment date that identified PD. If subject died without PD, PD date was death date. For surviving subjects who didn't have documented PD, DOR was censored at last radiologic assessment. For subjects who receive subsequent anti-cancer therapy prior to documented PD, DOR was censored at last radiologic assessment prior to commencement of subsequent therapy. Subjects who had an initial PD event immediately following 2 or more consecutive missed assessments were censored at last assessment prior to missed assessments. DOR was only calculated for subjects with a best response of PR or CR.
Time Frame: From date of first response to date of progression/death, or censored as described above; assessed for approximately 2 years.
Population: The evaluable population for efficacy includes subjects who receive initial placement of the NovoTTF100A transducer arrays. Note: 4 subjects discontinued study participation prior to device placement, and are therefore are excluded from efficacy analyses. Duration of response was conducted specifically on those subjects in the efficacy population who achieved objective response (PR or CR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Planned RT + TMZ + BEV + NovoTTF100A Device
Number analyzed (Participants) | 3
months | 8.1 [3.7 to 8.6]
Statistical Analysis 1: Comparison: Planned RT + TMZ + BEV + NovoTTF100A Device; Test type: Other — Estimation only; Median = 8.1, 95% CI 2-sided [3.7 to 8.6] — The Kaplan Meier method was used to estimate median duration of response (in months). The Greenwood method was used to estimate confidence limits of median duration of response

7. Secondary Outcome: Duration of Disease Control
Description: Duration of disease control (DoDC) was measured from the time of initiation of chemoradiation therapy until the first occurrence of either progressive disease or death. PD must be objectively determined as per RANO criteria (Updated Response Assessment Criteria for High Grade Gliomas, where PD is defined as a 25% increase in sum of products of diameters from nadir), where PD date is assessment date that identified PD. If subject died without PD, PD date was death date. For surviving subjects who didn't have documented PD, DoDC was censored at last radiologic assessment. For subjects who receive subsequent anti-cancer therapy prior to documented PD, DoDC was censored at last radiologic assessment prior to commencement of subsequent therapy. Subjects who had an initial PD event immediately following 2 or more consecutive missed assessments were censored at last assessment prior to missed assessments. DoDC was calculated only for subjects with a best overall response of SD or better.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Planned RT + TMZ + BEV + NovoTTF100A Device
Number analyzed (Participants) | 9
months | 7.9 [4.8 to 10.4]
Statistical Analysis 1: Comparison: Planned RT + TMZ + BEV + NovoTTF100A Device; Test type: Other — Estimation Only; Median = 7.9, 95% CI 2-sided [4.8 to 10.4] — The Kaplan Meier method was used to estimate median duration of disease control (in months). The Greenwood method was used to estimate confidence limits of median duration of disease control

ADVERSE EVENTS:
Time Frame: Baseline, during treatment [concurrent chemoradiation phase (6 weeks +/- 7 days, pre-NovoTTF100A system treatment (up to 2 weeks), NovoTTF100A system treatment with TMZ/BEV maintenance for up to 12 cycles], and through 30 days after NovoTTF100A device is discontinued or 30 days after last dose of study treatment for those who do not have NovoTTF100A device placed, up to approximately 66 weeks.
Arm/Group | Planned RT + TMZ + BEV + NovoTTF100A Device
All-Cause Mortality (participants affected / at risk) | 11/13
Serious Adverse Events (participants affected / at risk) | 8/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Planned RT + TMZ + BEV + NovoTTF100A Device (N=13)
Encephalopathy (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 2
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 — Lung infection
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Planned RT + TMZ + BEV + NovoTTF100A Device (N=13)
Fatigue (General disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 10
Fall (Injury, poisoning and procedural complications) | 9
Anorexia (Metabolism and nutrition disorders) | 8
Headache (Nervous system disorders) | 7
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7
Nausea (Gastrointestinal disorders) | 6
Platelet count decreased (Investigations) | 6
Confusion (Psychiatric disorders) | 5
Constipation (Gastrointestinal disorders) | 5
Dysgeusia (Nervous system disorders) | 5
Skin ulceration (Skin and subcutaneous tissue disorders) | 5
Depression (Psychiatric disorders) | 4
Gait disturbance (General disorders) | 4
Memory impairment (Nervous system disorders) | 4
Weight loss (Investigations) | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 4
Anxiety (Psychiatric disorders) | 3
Blurred vision (Eye disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Dysphasia (Nervous system disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Insomnia (Psychiatric disorders) | 3
Thromboembolic event (Vascular disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 3
Urinary tract infection (Infections and infestations) | 3
Localized edema (General disorders) | 3
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 3
Bloating (Gastrointestinal disorders) | 2
Bruising (Injury, poisoning and procedural complications) | 2
Cognitive disturbance (Nervous system disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Dizziness (Nervous system disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Encephalopathy (Nervous system disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Personality change (Psychiatric disorders) | 2
Photosensitivity (Skin and subcutaneous tissue disorders) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 — Pulmonary inflammation
Seizure (Nervous system disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Weight gain (Investigations) | 2
Facial muscle weakness (Nervous system disorders) | 2
Mucosal infection (Infections and infestations) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
Adrenal insufficiency (Endocrine disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Amnesia (Nervous system disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Cardiac disorders - Other (Cardiac disorders) | 1 — Left ventricular hypertrophy
CD4 lymphocytes decreased (Investigations) | 1
Chills (General disorders) | 1
Conjunctivitis (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Edema face (General disorders) | 1
Eye disorders - Other (Eye disorders) | 1 — Vision changes - intermittent
Fever (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Infections and infestations - Other (Infections and infestations) | 1 — Shingles
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 — Electric sensation scalp
Lethargy (Nervous system disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Malaise (General disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Paresthesia (Nervous system disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Psychosis (Psychiatric disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 — Dysuria
Restlessness (Psychiatric disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Skin infection (Infections and infestations) | 1
Somnolence (Nervous system disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Tremor (Nervous system disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary frequency (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal infection (Infections and infestations) | 1
Vaginal inflammation (Reproductive system and breast disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Watering eyes (Eye disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1
Edema limbs (General disorders) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — Skin erosion
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — Skin irritation
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — Skin tears
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 — Pinpoint non-petechial lesions to bilateral hands
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 — Lung infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-05): https://cdn.clinicaltrials.gov/large-docs/49/NCT02343549/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/49/NCT02343549/ICF_001.pdf